CLINICAL TRIAL: NCT06459466
Title: Effects of Kinesiotherapy Exercises Along With Cervical Mobilization in Cervicobrachial Neuralgia.
Brief Title: Effects of Kinesiotherapy Exercises With Cervical Mobilization in Cervicobrachial Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01116
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Cervico-Brachial Neuralgia
Keywords: kinesiotherapy; exercises; cervical mobilization
MeSH Terms: conditions — Brachial Plexus Neuritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotherapy exercises with cervical mobilization (Experimental): This group will receive kinesiotherapy exercises along with Cervical Mobilization
  Interventions: Procedure: kinesiotherapy exercises with cervical mobilization; Procedure: cervical Mobilization
- Cervical Mobilization (Active Comparator): This group will receive Cervical lateral glide mobilization.
  Interventions: Procedure: kinesiotherapy exercises with cervical mobilization; Procedure: cervical Mobilization

INTERVENTIONS:
Procedure: kinesiotherapy exercises with cervical mobilization — Kinesiotherapy Exercises includes Neck stretches , shoulder and upper back mobility, pectoral stretch, cervical isometrics, shoulder blade protraction and retraction
Procedure: cervical Mobilization — This includes Cervical lateral glide mobilization

SUMMARY:
To evaluate the effects of kinesiotherapy exercises with cervical mobilization in Cervicobrachial Neuralgia.

DETAILED DESCRIPTION:
Cervicobrachial Neuralgia is characterized by pain and discomfort in the arm, specifically in conjunction with pain in the cervical spine. It has been observed that a significant number of patients seeking therapy for cervical spine diseases are affected by this type of pain. When an illness is chronic, it has a tendency to manifest as a persistent or recurring issue that has a negative impact on an individual's mental and physical well-being.

It is a randomized clinical trial. 30 patients fulfilling the inclusion and exclusion criteria will be recruited by non-probability convenience sampling and then randomly divided in two groups using lottery method. Group A will receive the strengthening and kinesiotherapy exercises along with Brugger's relief position training with 10 minutes per session and cervical lateral glide mobilization, 3 times a week. And the group B will receive the cervical lateral glide mobilization. Pain levels will be measured using a visual analogue scale and goniometer will be used to measure neck ranges.The data will be analyzed by using SPSS version25.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age: 30-50 years
* Positive upper limb neurodynamic test
* Patients having neck pain radiating to upper limb and limited ROM with articular dysfunction.

Exclusion Criteria:

* Patients diagnosed with fibromyalgia
* Surgery of cervical/thoracic spine
* Limited glenohumeral joint movement
* Presence of neurological disease (stroke, multiple sclerosis)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain: Visual analogue scale (VAS) | 3 weeks
  VAS is a psychometric instrument used to measure subjective characteristics or attitudes, typically pain intensity or other subjective experiences.

SECONDARY OUTCOMES:
Range of Motion: Goniometer | 3 weeks
  It is an instrument used to measure angles, typically the range of motion of joints in the human body.

OTHER OUTCOMES:
Cervical radiculopathy impact scale (CRIS) | 3 weeks
  It is a 21-item self-reported questionnaire that is used to assess the impact of cervical radiculopathy on patients' daily lives. It is divided into three subscales:
  * Symptoms (9 items)
  * Energy and postures (6 items)
  * Actions and activities (6 items)

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- IIMCT Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rigal M, Portet S, Jouanneau E, Riva R, Eker O, Jacquesson T. Cervicobrachial neuralgia due to vertebral artery loop. Surg Radiol Anat. 2022 Feb;44(2):223-226. doi: 10.1007/s00276-022-02885-z. Epub 2022 Jan 23. PMID 35066610
- [Background] Gangavelli R, Nair NS, Bhat AK, Solomon JM. Cervicobrachial pain - How Often is it Neurogenic? J Clin Diagn Res. 2016 Mar;10(3):YC14-6. doi: 10.7860/JCDR/2016/16456.7492. Epub 2016 Mar 1. PMID 27134988
- [Background] Coudert P, Laine G, Pointillart V, Damade C, Boissiere L, Vital JM, Bouyer B, Gille O. Tomodensitometric bone anatomy of the intervertebral foramen of the lower cervical spine: measurements and comparison of foraminal volume in healthy individuals and patients suffering from cervicobrachial neuralgia due to foraminal stenosis. Surg Radiol Anat. 2022 Jun;44(6):883-890. doi: 10.1007/s00276-022-02941-8. Epub 2022 Apr 28. PMID 35477797
- [Background] Kouki S, Landolsi M, Ben Lassoued M, Gharsallah I. Uncommon cause of cervicobrachial neuralgia: epidural abscess complicating tuberculous arthritis. BMJ Case Rep. 2017 Jul 17;2017:bcr2017219458. doi: 10.1136/bcr-2017-219458. No abstract available. PMID 28716773
- [Background] Mostofi K, Peyravi M, Moghadam BG. Cervicothoracic junction disc herniation: Our experience, technical remarks, and outcome. J Craniovertebr Junction Spine. 2020 Jan-Mar;11(1):22-25. doi: 10.4103/jcvjs.JCVJS_102_19. Epub 2020 Apr 4. PMID 32549708
- [Background] Thoomes E, Ellis R, Dilley A, Falla D, Thoomes-de Graaf M. Excursion of the median nerve during a contra-lateral cervical lateral glide movement in people with and without cervical radiculopathy. Musculoskelet Sci Pract. 2021 Apr;52:102349. doi: 10.1016/j.msksp.2021.102349. Epub 2021 Feb 16. PMID 33618231
- [Background] Huber J, Lisinski P, Polowczyk A. Reinvestigation of the dysfunction in neck and shoulder girdle muscles as the reason of cervicogenic headache among office workers. Disabil Rehabil. 2013 May;35(10):793-802. doi: 10.3109/09638288.2012.709306. Epub 2012 Aug 14. PMID 22888759
- [Background] Martin-Vera D, Fernandez-Carnero J, Rodriguez-Sanz D, Calvo-Lobo C, Lopez-de-Uralde-Villanueva I, Arribas-Romano A, Martinez-Lozano P, Pecos-Martin D. Median Nerve Neural Mobilization Adds No Additional Benefit When Combined with Cervical Lateral Glide in the Treatment of Neck Pain: A Randomized Clinical Trial. J Clin Med. 2021 Nov 5;10(21):5178. doi: 10.3390/jcm10215178. PMID 34768696